CLINICAL TRIAL: NCT01861691
Title: Randomized Controlled Trial to Evaluate Laparoscopic Versus Open Surgery in Transverse and Descending Colon Cancer Patients
Brief Title: Randomized Controlled Trial Between Laparoscopic and Open Surgery in Transverse and Descending Colon Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shoichi Fujii, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Shoichi Fujii, MD, PhD, Associate Professor, Yokohama City University Medical Center
Organization: Yokohama City University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YCUMC-D1108014; YokohamaCUMC33 (Other: YokohamaCUMC)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Malignant Neoplasm of Transverse Colon; Malignant Neoplasm of Descending Colon
Keywords: Transverse colon cancer; Descending colon cancer; Laparoscopic surgery; Randomized controlled trial
MeSH Terms: interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open surgery (Active Comparator): Open colectomy
  Interventions: Procedure: Open surgery
- Laparoscopic surgery (Experimental): Laparoscopic colectomy
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Open surgery — Conventional technique
  Other Names: Open colectomy
  Arms: Open surgery
Procedure: Laparoscopic surgery — New minimum invasive technique
  Other Names: Laparoscopic colectomy
  Arms: Laparoscopic surgery

SUMMARY:
The long-term results of several large-scale prospective randomized trials that compared laparoscopic-assisted and open colectomy for colon cancer were published in the past decade. The oncologic outcomes were nearly similar in patients who underwent laparoscopic or open surgery. In Japan, the Japan Clinical Oncology Group (JCOG) conducted a randomized trial to compare oncological outcomes between patients who underwent laparoscopic or open surgery for advanced colon cancer and recto-sigmoid cancer. However, the exclusion criterion were concerning tumor site in transverse and descending colon. The reason of exclusion was that laparoscopic procedure was difficult in transverse and descending colon cancers. However, laparoscopic surgery for transverse and descending colon cancer was performed clinically. We conducted a randomized trial that compared laparoscopic surgery and conventional open surgery in in transverse and descending colon cancer. The purpose of the present study was to clarify the safety and feasibility of laparoscopic surgery on in transverse and descending colon cancer patients.

DETAILED DESCRIPTION:
Patients

* This was a randomized controlled trial conducted at a single institute, which was Yokohama City University Medical Center (Japan).
* 80 patients who had transverse colon or descending colon cancer were randomly allocated to receive laparoscopic surgery or conventional open surgery.

Surgical procedures

* All surgical procedures were performed by one specialized colorectal treatment team. The laparoscopic surgeries were performed by a surgeon who passed the skill accreditation system for laparoscopic gastroenterological surgery was established by the Japanese Society for Endoscopic Surgery (JSES), and all open surgeries were performed under the supervision of these skillful surgeons.
* All operations were performed according to the standard radical cure procedure described in the seventh edition of the Japanese General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus. That is, intestinal excision with lymph node dissection that separated the feeding blood vessel at its origin was performed in all surgical procedures. Patients who underwent palliative partial excision were not included.
* In the laparoscopic surgery, a medial-to-lateral approach was performed in all patients.
* In the conventional open surgery, the first procedure was done in lateral approach. The reconstruction techniques were the same as those used in laparoscopic surgery.

Randomization - To balance the operative backgrounds between the laparoscopic and the conventional open surgery groups, the patients were stratified by the tumor location (transverse colon, descending colon).

Adjuvant therapy

* When the pathological stage was diagnosed as stage 3 by histological examination of the resected specimen, adjuvant chemotherapy was done with oral fluoropyrimidine anti-cancer drug.
* Neither radiation therapy nor preoperative chemotherapy was given to any patient. Preoperative chemo-radiotherapy even for rectal cancer is not yet standard treatment in Japan.

Assessment parameters

* The preoperative parameters
* Operative assessment parameters
* Postoperative assessment parameters An early postoperative complication was defined as a complication that occurred between the finish of the operation and postoperative day 30. A late postoperative complication was defined as a complication that occurred after postoperative day 30. The terminologies of complications were classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and grading was done by Classification of Surgical Complication.
* The pathological results were recorded according to the 7th edition of the Japanese General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus and 7th edition of primary tumor, regional nodes, metastasis (TNM) classification. Circumferential margin involvement was defined as exposure of a cancer cell at the vertical dissection surface on histological examination.
* Quality of life (QOL) scores. The QOL score was measured using the 36-item Short Form Health Survey (SF-36) version 2.0. It is a tool that measures health-related QOL (HRQOL) according to an inclusive standard and not a disease-specific standard. The SF-36 is composed of 36 questions. The score is expressed numerically by the provided scoring algorithm. SF-36 questionnaires were sent to the patients at one month, 6 months and one year after the surgery by postal mail. A return envelope was enclosed with the SF-36 questionnaire, and the patient sent it back to the research secretariat by postal mail. A questionnaire on the defecation situation and wound pain besides the SF-36 was added all three times. The question of when complete rehabilitation occurred was added in the questionnaire at one year.

Follow-up schedule

- The follow-up schedule was as follows according to stage. Patients with stages 0 and I were followed up with outpatient examinations including tumor marker measurements, and chest, abdominal and pelvic computed tomography (CT) once a year for five years. Patients with stage 2 and 3a were examined by CT and tumor marker measurements every six months for the first two years. These examinations were done once a year from the third year to the fifth year. Patients with stage 3b and 3c were examined by CT and tumor marker measurements every four months for the first two years, and every six months from the third year to the fifth year.

Statistical analysis

* The primary endpoint was early complication rate.
* The secondary endpoints were 5-recurrence-free survival, 5-year overall survival, length of postoperative hospital stay, and HRQOL score. To evaluate whether a difference in the operative procedure influences survival including death due to another disease, a comparison of overall survival has meaning. Early complication rate, length of postoperative hospital stay and HRQOL score were added to the secondary endpoints because these parameters had a possibility of becoming grounds of selection of the operation method if there were no differences in overall survival and recurrence-free survival.
* A sample size of 74 patients was assured to achieve a power of more than 70% to detect a difference between the groups using a two-sided Chi-squared test with type I error rate equal to 0.2, when the true complication rates were 20% and 40% for the laparoscopic and open surgeries, respectively. The dropouts were considered and the number of accumulation targets was assumed to be 80 patients.
* For continuous variables, data are presented as means ± standard deviation (SD). For categorical variables, data are presented as frequencies and percentages (%). Comparison of the endpoints was based on intention-to-treat principle, that is, the patients who switched to another group during surgery were treated as members of the allocated group. The Chi-squared test was applied to evaluate the significance of differences in proportions, and t-test was used to evaluate the significance of differences in continuous variables. A p-value of less than 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age of 20 years old or over
* Histologically proven adenocarcinoma
* Clinical tumor penetrates visceral peritoneum (T4a), no metastasis (M0) or lower T factor
* Elective operation
* Tolerable surgery under general anesthesia
* No bulky tumor larger than 8cm in diameter
* No history of laparotomy for colorectal resection except appendectomy
* Provided written informed consent

Exclusion Criteria:

* Synchronous or metachronous (within 5 years) malignancy in another organ except carcinoma in situ
* Multiple colorectal cancer that needs reconstruction two or more times
* Acute intestinal obstruction or perforation due to colorectal cancer
* Lower rectal cancer that required pelvic side wall lymphadenectomy
* Pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-08; Primary Completion 2012-10 (Actual); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Early complication rate | within the first 30 days after surgery
  Early complication is defined as a complication that occured between the finish of the surgery and postoperative day 30.

SECONDARY OUTCOMES:
Recurrence-free survival | 5 years
  All death and recurrence of colon cancer is defined as an event of recurrence-free survival.
Overall survival | 5 years
  All death is defined as an event of overall survival.
Length of postoperative hospital stay | 10 days
  Length of postoperative hospital stay is defined as a duration between surgery and first discharge. An expected average is 10 days.
Health-related QOL score | 1 year after surgery
  The QOL score was measured using the 36-item Short Form Health Survey (SF-36) version 2.0. It is a tool that measures health-related QOL (HRQOL) according to an inclusive standard and not a disease-specific standard. The SF-36 is composed of 36 questions. The score is expressed numerically by the provided scoring algorithm. SF-36 questionnaires were sent to the patients at one month, 6 months and one year after the surgery by postal mail. A return envelope was enclosed with the SF-36 questionnaire, and the patient sent it back to the research secretariat by postal mail. A questionnaire on the defecation situation and wound pain besides the SF-36 was added all three times. The question of when complete rehabilitation occurred was added in the questionnaire at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Chikara Kunisaki, Professor, Study Chair — Yokohama City University, Gastroenterological Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan

REFERENCES:
- [Derived] Toritani K, Watanabe J, Nakagawa K, Suwa Y, Suwa H, Ishibe A, Ota M, Fujii S, Kunisaki C, Endo I. Randomized controlled trial to evaluate laparoscopic versus open surgery in transverse and descending colon cancer patients. Int J Colorectal Dis. 2019 Jul;34(7):1211-1220. doi: 10.1007/s00384-019-03305-2. Epub 2019 May 17. PMID 31102008